CLINICAL TRIAL: NCT00256035
Title: IL-4 as a Marker of Atherosclerosis
Brief Title: Interleukin-4 (IL-4) as a Marker of Atherosclerosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Melbourne Health (Other)
Collaborators: The Intensive Care Unit Departmental Funding (Unknown)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2002.156
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Atherosclerosis; Ischemic Heart Disease
MeSH Terms: conditions — Atherosclerosis; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Unstable coronary artery disease (Other): Patients with unstable coronary artery disease will have daily IL6 levels
  Interventions: Procedure: Measuring IL-4 levels
- Coronary Angioplasty Patients (Other): Patients having coronary angioplasty will have levels taken before and immediately after the proceedure and 24 hours post.
  Interventions: Procedure: Measuring IL-4 levels
- Coronary bypass grafts patients (Other): Patients will have levels collected immediately after and 24 hours post procedure
  Interventions: Procedure: Measuring IL-4 levels
- Stable coronary Artery Diseaese Patients (Other): Once the patients are commenced on treatment with statins and or angiotensin converting enzyme they will have twice weekly levels taken
  Interventions: Procedure: Measuring IL-4 levels

INTERVENTIONS:
Procedure: Measuring IL-4 levels

SUMMARY:
In recent years, medical research into the cause and progression of heart disease due to narrowing and blockage of blood vessels to the heart muscle has improved the understanding of ischemic heart disease. It is now accepted that both the development and later progression with sudden blockage of blood vessels are associated with inflammation, although it remains unknown exactly what triggers this inflammatory process. It is possible that new blood tests which measure markers of inflammation in the bloodstream may be useful to help identify patients at risk of heart damage and assess response to treatment.

The study plans to assess a new blood test for a known marker of inflammation (IL-4) in patients with heart disease.

The hypothesis of this study is that, the cytokine, IL-4, measured by a new assay, is abnormally elevated in the blood of patients with coronary artery disease.

Also hypothesized is that the degree of abnormality of blood IL-4, is related to important clinical events in such patients, including severity of disease, acute complications, and treatment.

DETAILED DESCRIPTION:
This is a single centre, prospective, non randomised, non controlled, pilot study of the potential abnormality of a new test group of patients in whom the results are postulated to be abnormal.

The specific aims of the study are:

1. To measure IL-4 by a new rapid on-site technique in patients with documented coronary artery disease presenting in a variety of acute clinical circumstances
2. To evaluate any abnormal measurements in relation to the severity of the disease, acute vascular complication and newly prescribed medications.

It is proposed to study 4 small groups of patients with ischemic heart disease.

1. Patients with unstable coronary artery disease admitted to the Coronary Care Unit. They will be studied on admission and then daily until coronary angiography is performed.
2. Patients having coronary angioplasty. They will be studied before, immediately after and 24 hours after the procedure.
3. Patients having coronary artery bypass grafting will be studied immediately after and 24 hours post surgery.
4. Patients with stable coronary artery disease about to receive a statin and or angiotensin-converting enzyme inhibitor therapy will be studied before and twice weekly after commencement of therapy for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All patients (either sex and any age) presenting in the settings described will be eligible to participate.

Exclusion Criteria:

* An unwillingness to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To measure the IL-4 by a new rapid point-of-care technique in patients with documented coronary artery disease presenting in a variety of acute clinical circumstances | Hospital Discharge

SECONDARY OUTCOMES:
To evaluate any abnormal measurements in relation to the severity of the disease, acute vascular complications, and newly prescribed medications | Hospital Discharge

CONTACTS AND LOCATIONS:
Overall Officials: Megan Robertson, Principal Investigator — Melbourne Health